CLINICAL TRIAL: NCT00623285
Title: The Effects of Peri-operative Pregabalin Administration on Post-operative Analgesia in Patients Undergoing Coronary Bypass Grafting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Joel Loiselle, MD, FRCPC, St. Boniface General Hospital/University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG2007; AOC
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Pain.
Keywords: Pain.; Postoperative.; CABG.
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Pregabalin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Pregabalin
- Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo/Lactose

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150mg orally 60 minutes pre-operatively. Patients will receive the first dose post-operatively 12 hours after the initial dose was taken (+ 6 hours) given that patient is able to swallow and then they will receive 150mg twice a day through the first 2 post-operative days for a total of six doses.
  Other Names: Lyrica
  Arms: Group 1
Drug: Placebo/Lactose — Matching Placebo orally,60 minutes pre-operatively. Patients will receive the first dose post-operatively 12 hours after the initial dose was taken (+ 6 hours) given that patient is able to swallow and then they will receive placebo twice a day through the first 2 post-operative days for a total of six doses. If the patient is unable to swallow and NG tube is in place, the medication can be dissolved in water and administered through the NG tube.
  Arms: Group 2

SUMMARY:
We hypothesize that the perioperative administration of pregabalin will significantly decrease pain scores and post-operative opioid requirements for patients undergoing coronary artery bypass grafting, and reduces the incidence of opioid-induced side effects such as respiratory depression. This may reduce ICU admission and possibly abbreviate length of hospital stay.

ELIGIBILITY:
Inclusion Criteria

* Patients whom are able and willing to provide written informed consent.
* Male and female 18-70 years of age.
* Patients whom are undergoing isolated coronary artery bypass grafting through a midline sternotomy for the treatment of ischemic heart disease.

Exclusion criteria

* Patients undergoing cardiac surgery for valvular or pericardial surgery.
* Patients with a documented ejection fraction of less than 50%.
* Patients with known chronic renal insufficiency and a calculated creatinine clearance of < 60mL/min.
* Patients with known sensitivity to the study drugs.
* Patients with documented pre-existing chronic pain.
* Patients with seizure disorders.
* Patients whom are taking pregabalin or gabapentin
* Patients on chronic neuroleptic medications for control of psychiatric disorders as to avoid possible drug interactions and to avoid modulation of any pain states by such medications.
* Patients whom are taking tricyclic antidepressants or serotonin and norepinephrine re-uptake inhibitors(SNRI) will be excluded because of the effect of these drugs on neuropathic pain.
* Patients greater than 70 years of age will also be excluded because of their increased risk of side-effects and perioperative confusion.
* Pregnant or breast feeding females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Pain scores and morphine consumption post surgery | 6 months

SECONDARY OUTCOMES:
To determine the occurrence of opioid-related side effects such as nausea, vomiting, and respiratory depression in patients receiving pregabalin compared to those receiving placebo. | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Loieselle, MD, Principal Investigator — St. Boniface General Hospital and U of M
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada